CLINICAL TRIAL: NCT02302664
Title: A Pragmatic Multi-centre Blinded Randomised Placebo-controlled Trial Comparing Platelet Rich Plasma Injection (PRP) to Placebo (Imitation) Injection in Adults With Achilles Tendon Rupture
Brief Title: PATH-2: Platelet Rich Plasma in Achilles Tendon Healing
Acronym: PATH-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14/SC/1333
Record Dates: First submitted 2014-11-18; First posted 2014-11-27 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2017-06

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles; Platelet Rich Plasma; Patient reported outcome measure; Orthopaedic trauma; Musculoskeletal; Tendon; Sports Injury; Heel-Rise Endurance Test
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP Injection (Active Comparator): Intervention - PRP Injection: The injection is the intervention. A blood sample is withdrawn from patient. Away from patient part of sample is spun down in centrifuge to produce 'Platelet Rich Plasma' (PRP). Patient returns to treatment area and their own PRP is then injected into tendon rupture gap. This is carried out by a surgeon or extended scope physiotherapist, generally in the outpatient clinic, after a local anaesthetic has been applied. Patient is lying face down during procedure, unaware of treatment given to tendon at back of leg. Remaining blood sample sent for analysis.
  Interventions: Procedure: PRP Injection into Achilles tendon rupture gap
- Imitation Injection (Sham Comparator): Sham - Imitation Injection: The injection is the intervention. A blood sample is withdrawn from patient. Treatment is prepared. Patient returns to treatment area and a needle (no syringe) is inserted and held into tendon rupture gap to mimic injection (after local anaesthetic has been applied). No active ingredient given. Carried out by surgeon or extended scope physiotherapist, generally in the outpatient clinic. Patient is lying face down during procedure, unaware of treatment given to tendon at back of leg. Blood sample sent for analysis.
  Interventions: Procedure: Imitation Injection into Achilles tendon rupture gap

INTERVENTIONS:
Procedure: PRP Injection into Achilles tendon rupture gap — PRP injection delivered into the tendon rupture gap Intervention - PRP Injection: The injection is the intervention. A blood sample is withdrawn from patient. Away from patient part of sample is spun down in centrifuge to produce 'Platelet Rich Plasma' (PRP). Patient returns to treatment area and their own PRP is then injected into tendon rupture gap. This is carried out by a surgeon or extended scope physiotherapist, generally in the outpatient clinic, after a local anaesthetic has been applied. Patient is lying face down during procedure, unaware of treatment given to tendon at back of leg. Remaining blood sample sent for analysis.
  Arms: PRP Injection
Procedure: Imitation Injection into Achilles tendon rupture gap — Imitation injection delivered into the tendon rupture gap Sham - Imitation Injection: The injection is the intervention. A blood sample is withdrawn from patient. Treatment is prepared. Patient returns to treatment area and a needle (no syringe) is inserted and held into tendon rupture gap to mimic injection (after local anaesthetic has been applied). No active ingredient given. Carried out by surgeon or extended scope physiotherapist, generally in the outpatient clinic. Patient is lying face down during procedure, unaware of treatment given to tendon at back of leg. Blood sample sent for analysis.
  Arms: Imitation Injection

SUMMARY:
Platelet Rich Plasma in Achilles Tendon Healing

Does using a Platelet Rich Plasma (PRP) injection immediately before standard casting benefit patients aged 18 or over who are suitable for nonsurgical treatment of the Achilles tendon rupture (ATR)? This is a multicentre, blinded, randomised, placebo controlled trial with two sub studies: (1) blood sample analysis and (2) needle biopsy in 16 participants.

ATR is the most common tendon injury and leads to months of incapacity. With an average work absence of 63108 days there are significant societal and National Health Service (NHS) costs. PRP potential benefit is to improve recovery and return to normal activities earlier, and reduce the NHS and societal impact. The investigators will investigate the efficacy of PRP using disease specific and patient important outcomes to improve the evidence for this treatment of ATR.

A minimum of 15 United Kingdom (UK) NHS hospitals will be included to recruit 214 participants. Patients will be identified in the orthopaedic outpatient clinic, usually following an emergency hospital attendance for ATR. After checking eligibility and the informed consent process, baseline data is collected and participants randomised to either 'PRP injection' or 'Imitation (placebo) injection'. A participant's own blood sample is taken and prepared according to allocation. The injection is delivered by a trained surgeon in clinic who will be aware of allocation while the participant remains blind.

Participants complete a pain diary and have four study assessments at 4,7,13 and 24 weeks, carried out by a member of the research team blind to allocation. Assessments take place over the telephone or during a hospital outpatient visit. The 24 week hospital visit includes an exercise test of ankle function. All assessments include collection of patient reported responses to pre-set questions.

The results may be applicable to the many other tendon and ligament injuries. The National Institute for Health Research (NIHR)/Medical Research Council (MRC) Efficacy and Mechanism Evaluation Programme provides funding and University of Oxford is Sponsor.

DETAILED DESCRIPTION:
PURPOSE The aim of this study is to evaluate the effectiveness of treating ruptured Achilles tendon with autologous platelet rich plasma. The investigators plan to compare the outcome of traditional methods of immobilisation in a cast with the outcome of the same methods after applying platelet rich plasma to the ruptured tendon.

Spontaneous rupture of the Achilles tendon is the most common tendon injury in the human body, it accounts for approximately 20% of all major tendon ruptures. Since the 1950s, the incidence of Achilles tendon rupture has been increasing. The peak incidence of ATR is between 30 and 40 years of age. Current treatments are associated with a significant risk of rerupture for the Achilles tendon; this is up to 15%. Therapies are currently dominated by the conflicting priorities of rapid rehabilitation and a return to work versus the risk of rerupture and/or surgery. New cost effective treatments that reduce both the risk of rerupture and time to functional healing are needed to address this challenge.

Platelets are blood cells that form blood clots in the injured tissues. Platelets have evolved over millennia to deliver a combinatorial wound healing cocktail that comprises over 1100 active soluble and membrane bound components, delivered sequentially over a timeframe from minutes to the lifespan of the platelets. Platelets and platelet derived growth factors play important roles in the healthy response to injury, promoting healing of tissues, and have been proposed as therapeutic agents. Their potential for tendon repair has been demonstrated in laboratory experiments and animal models. One human investigation has been published, a small study in athletes showing accelerated return to function with platelet preparations from patients own blood after complete Achilles tendon rupture. However, there has been no scientifically sound clinical research to assess the full potential of using platelet preparations to accelerate healing of Achilles tendon.

Despite that lack of high quality trial data, PRP administration remains a potentially attractive strategy to explore given it is of relatively low cost and minimally invasive. There has been a recent steep growth in PRP use for musculoskeletal conditions. It is estimated that PRP is used to treat 86,000 tendon disorders annually in the United States and a similar number in Europe.

There is also evidence that PRP injections are being introduced in NHS clinical practice, in addition to a wider use in private medicine within the United Kingdom. The investigators surveyed the declarations of use of PRP in NHS hospitals and discovered four offering PRP for tendon injuries. Without evidence of efficacy the consequences range from the NHS incurring extra costs for a treatment with unproven clinical effects to the non deployment of an effective autologous intervention. There is therefore a pressing need to undertake this study before the use of PRP becomes widely adopted. The results of this study may inform the design of a potential future clinical trial of optimal PRP therapy versus surgical repair for ATR in restoring patient function.

The National Institute for Health and Care Excellence (NICE) review of PRP use (IPG 438) states that specialist advisers noted that this was an established practice and it is of concern that participants are being exposed to these intervention techniques without adequate clinical investigation into their efficacy and validity. NICE encourages further research comparing autologous blood injections (with or without techniques to produce PRP) against established nonsurgical methods.

The proposed trial aims are:

1. Evaluate the clinical efficacy of PRP in acute ATR in terms of mechanical muscle tendon function.
2. Evaluate the clinical efficacy of PRP in acute ATR in terms of patient reported functional recovery, pain and quality of life.
3. Determine the key components of PRP that contribute to its mechanism of action.
4. Explore the immunohistochemical response of the healing tendon to PRP at the cellular and tissue level.

STUDY DESIGN Platelet Rich Plasma in Achilles Tendon Healing (PATH-2) is a pragmatic prospective multicentre, blinded, randomised, placebo controlled trial with two sub studies embedded within the main study. The study aims to evaluate the clinical efficacy of PRP in acute ATR in terms of mechanical muscle tendon function. To achieve the goals of this study and produce high level evidence of PRP efficacy, the study is a randomised controlled trial. The randomisation will reduce the risk of bias and the control arm will help to eliminate the placebo effect. Patients and assessors are blinded to the applied treatment to reduce the risk of bias.

The PATH-2 study will take place in a minimum of 15 NHS hospitals across the UK. Participants will be identified in the orthopaedic/trauma outpatient clinic, usually following an emergency hospital attendance for an Achilles tendon rupture. The investigators anticipate the surgeon will confirm appropriateness for nonsurgical treatment and eligibility. A member of the local research team will carry out the informed consent process, baseline data collection and randomisation.

Participants will be randomised via a telephone or website randomisation service, and will be allocated to receive either 'PRP injection' or 'Imitation (placebo) injection'. Treatment will be administered by a surgeon during the outpatient visit. Those involved in treatment delivery will be aware of treatment allocation due to the nature of the intervention. Participants should remain blind to allocation throughout the study.

There are blinded outcome assessments at 4, 7, 13 and 24 weeks and 24 months after treatment. For the first three (4, 7, 13 weeks) responses will be collected over the telephone or during a hospital outpatient visit (where this coincides with local follow-up). The fourth follow-up requires a hospital attendance at 24 weeks, with a face-to-face interview and assessment by a physiotherapist/assessor. At this visit, the primary outcome (HRET) will be collected. The final follow-up (24 months) is completed by post or telephone.

The two embedded sub studies are:

1. Sub study 1: Blood component (all participants, all sites) and PRP component analyses (PRP intervention arm only). A blood sample will be taken from each participant after consent and randomisation but prior to treatment. The samples will be analysed to compare its composition by blood cell type. PRP samples will be prepared according to treatment allocation and a portion will remain after treatment. This will be sent to a central laboratory for later analysis (blood cells count, growth factors and platelets viability).
2. Sub study 2: Immunohistochemistry analysis (16 participants from selected sites only who have given consent to undergo the sample collection procedure). A needle biopsy of the healing Achilles tendon under ultrasound guidance will be taking during an outpatient visit. Samples will undergo immunohistochemistry analysis centrally in a specialist laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to give informed consent for participation in the study
* Aged 18 years or over
* Ambulatory prior to injury without the use of walking aids or assistance of another person
* Diagnosed with an acute, complete, Achilles tendon rupture
* Presenting within and receiving study treatment within 12 days post injury
* Patients in whom the decision has been made for non-operative treatment
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Able to attend a PATH-2 study hospital site for the 24-week follow-up.

Exclusion Criteria:

The patient may not enter the study if any of the following apply:

* Achilles tendon injuries at the insertion to the calcaneum or at the musculotendinous junction
* Previous major tendon or ankle injury or deformity to either lower leg
* History of diabetes mellitus
* Known platelet abnormality or haematological disorder
* Current use of systemic cortisone or a treatment dose of an anticoagulant (i.e. a prophylactic dose for preventing thrombosis would not be an exclusion)
* Evidence of lower limb gangrene/ulcers or peripheral vascular disease
* History of hepatic or renal impairment or dialysis
* Female patients who are pregnant or breast feeding
* Is currently receiving or has received radiation or chemotherapy within the last 3 months
* Has inadequate venous access for drawing blood
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Heel-Rise Endurance Test (HRET) | 24 weeks following study treatment
  Muscle-tendon function, measured objectively with the limb symmetry index (LSI) in maximal work during the heel-rise endurance test (HRET) [ Time Frame: 24 weeks following study treatment ] The HRET is a validated objective performant test of calf-muscle Achilles tendon capacity to work, which is measured in the unit joules (J). The HRET involves the participant standing on one leg and raising and lowering the heel repeatedly until fatigued. The work during the HRET for each lower limb is measured. The performance of each limb is then converted into a limb symmetry index, which is the primary outcome metric from the HRET.

SECONDARY OUTCOMES:
Number of heel rise repetitions | 24 weeks following study treatment
  Number of heel rise repetitions during the Heel-rise Endurance Test
Maximum heel rise height | 24 weeks following study treatment
  Maximum heel rise height (cm) during the Heel-rise Endurance Test
Achilles Tendon Rupture Score (ATRS) | 4, 7, 13 and 24 weeks and 24 months following study treatment
  Patient-report outcome measure (via questionnaire)
Patient Specific Functional Scale (PSFS) | 4, 7, 13, and 24 weeks and 24 months following study treatment
  Patient-report outcome measure (via questionnaire)
Short Form (SF-12 acute version) | 4, 7, 13, and 24 weeks and 24 months following study treatment
  Patient-report outcome measure (via questionnaire)
Pain diary - Visual analogue score (VAS) | 0-2 weeks following study treatment
  Daily pain diary

CONTACTS AND LOCATIONS:
Overall Officials: Keith Willett, Professor, Study Chair — Professor of Orthopaedic Surgery University of Oxford
Locations (18):
- United Kingdom (18):
  - John Radcliffe Hospital, Oxford, Oxford, Oxfordshire
  - Basildon University Hospital, Basildon
  - Southmead Hospital, Bristol
  - University Hospital of Wales, Cardiff
  - University Hospital Coventry, Coventry
  - Leighton Hospital, Crewe
  - Royal Devon & Exeter Hospital, Exeter
  - Royal Surrey Hospital, Guildford
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Aintree Hospital, Liverpool
  - Royal London Hospital, London
  - University Hospital South Manchester, Manchester
  - Peterborough City Hospital, Peterborough
  - Northern General Hospital, Sheffield
  - Morriston Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - Warrington & Halton Hospitals Trust, Warrington

REFERENCES:
- [Background] Keene DJ, Alsousou J, Willett K. How effective are platelet rich plasma injections in treating musculoskeletal soft tissue injuries? BMJ. 2016 Feb 17;352:i517. doi: 10.1136/bmj.i517. No abstract available. PMID 26888826
- [Derived] Schlussel MM, Keene DJ, Wagland S, Alsousou J, Lamb SE, Willett K, Dutton SJ; PATH-2 Trial Study Group. Platelet-rich plasma in Achilles tendon healing 2 (PATH-2) trial: statistical analysis plan for a multicentre, double-blinded, parallel-group, placebo-controlled randomised clinical trial. Trials. 2018 Aug 29;19(1):464. doi: 10.1186/s13063-018-2840-z. PMID 30157940
- [Derived] Alsousou J, Keene DJ, Hulley PA, Harrison P, Wagland S, Byrne C, Schlussel MM, Dutton SJ, Lamb SE, Willett K. Platelet rich Plasma in Achilles Tendon Healing 2 (PATH-2) trial: protocol for a multicentre, participant and assessor-blinded, parallel-group randomised clinical trial comparing platelet-rich plasma (PRP) injection versus placebo injection for Achilles tendon rupture. BMJ Open. 2017 Nov 16;7(11):e018135. doi: 10.1136/bmjopen-2017-018135. PMID 29150470